CLINICAL TRIAL: NCT01558102
Title: International Retrospective Study of Pipeline Embolization Device
Acronym: IntrePED
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: PED001
Record Dates: First submitted 2012-03-08; First posted 2012-03-20 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Brain Aneurysms
Keywords: brain aneurysm PED Pipeline
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this retrospective study is to determine the incidence of important safety outcomes in patients who have undergone Pipeline Embolization Device placement for intracranial aneurysms (IAs). This study does not effect patient care, simply it is designed to observe and capture information from numerous hospitals.

Data collection will be initiated starting March 2012 and continue until approximately April 2017.

ELIGIBILITY:
Inclusion Criteria:

* A patient who was treated with the Pipeline Embolization Device for treatment of a brain aneurysm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with brain aneurysms who were treated with the Pipeline Embolization Device
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Relative incidence of neurologic clinical events that occurred after treatment with PED | From Approval of PED in country of use until IRB approval at facility allowing for approximately 8-12 months of data for each subject. Outcomes are expected to be reported on 6 mo, 12mo, 2 yr, & 5yr data.
  Incidence of neurologic events from the time of Approval of the Pipeline Embolization Device in the country of use until IRB approval at facility.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Rush University Hospital, Chicago, Illinois
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Buffalo Neurosurgery, Buffalo General Hospital, Buffalo, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Fort Sanders Regional Medical Center, Neurovascular Research, Knoxville, Tennessee
- Clínica La Sagrada Familia, Buenos Aires, Argentina
- Royal University Hospital, Saskatoon, Saskatchewan, Canada
- Hôpital Gui de Chauliac, Montpellier, France
- National Institute of Neurosciences, Budapest, Hungary
- A.O. Ospedale Niguarda Ca' Granda, Milan, Italy

REFERENCES:
- [Derived] Park MS, Kilburg C, Taussky P, Albuquerque FC, Kallmes DF, Levy EI, Jabbour P, Szikora I, Boccardi E, Hanel RA, Bonafe A, McDougall CG. Pipeline Embolization Device with or without Adjunctive Coil Embolization: Analysis of Complications from the IntrePED Registry. AJNR Am J Neuroradiol. 2016 Jun;37(6):1127-31. doi: 10.3174/ajnr.A4678. Epub 2016 Jan 14. PMID 26767709